CLINICAL TRIAL: NCT06625723
Title: Investigating the Impact of a Sleep Aid on Sleep and Recovery Following Rotator Cuff Repair Surgery
Brief Title: Analysis of Sleep & Recovery Following Rotator Cuff Repair Surgery
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: New York Presbyterian Hospital (Other)
Responsible Party: Principal Investigator, Cole Morrissette, Resident Orthopedic Surgeon, New York Presbyterian Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ColumbiaOrthopedics
Record Dates: First submitted 2024-08-27; First posted 2024-10-03 (Actual); Last update posted 2024-11-18 (Actual); Status verified 2024-10

CONDITIONS: Rotator Cuff Tears; Rotator Cuff Injuries; Shoulder Pain; Shoulder Injuries; Shoulder Impingement
MeSH Terms: conditions — Rotator Cuff Injuries; Shoulder Pain; Shoulder Injuries; Shoulder Impingement Syndrome

STUDY DESIGN:
Intervention Model Description: Two treatment arms, one standard postoperative protocol following rotator cuff repair surgery. The second arm with the same protocol, with the addition of the sleep assistive device.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control Group (Active Comparator): Standard postoperative care for patients undergoing rotator cuff repair.
  Interventions: Procedure: Standard postoperative care
- Sleep Aid Group (Experimental): Standard postoperative care for patients undergoing rotator cuff repair PLUS the use of the sleep assistive device postoperatively.
  Interventions: Procedure: Standard postoperative care; Device: Surgical Recovery Systems Sleep Aid

INTERVENTIONS:
Procedure: Standard postoperative care — This will include medications, rehabilitation schedules, and follow-up visits as normally scheduled.
Device: Surgical Recovery Systems Sleep Aid — Sleep assistive device
  Arms: Sleep Aid Group

SUMMARY:
Postoperative recovery following a rotator cuff repair surgery can be challenging. In particular, sleeping is difficult given the restrictions of the operative shoulder. This study aims to evaluate a postoperative sleep device that will allow for safe and comfortable positioning of the arm, with the anticipated effect to improve postoperative recovery and sleep.

DETAILED DESCRIPTION:
Postoperative recovery following a rotator cuff repair surgery can be challenging. In particular, sleeping is difficult given the restrictions of the operative shoulder. This study aims to evaluate a postoperative sleep device that will allow for safe and comfortable positioning of the arm, with the anticipated effect to improve postoperative recovery and sleep.

ELIGIBILITY:
Inclusion Criteria:

* Rotator Cuff Tear

Exclusion Criteria:

* Prior ipsilateral shoulder surgery
* Ipsilateral upper extremity neurological deficit

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2026-10-01 (Estimated); Study Completion 2027-04-01 (Estimated)

PRIMARY OUTCOMES:
Narcotic Use | Daily
  Total amount of daily narcotics consumed for pain control.
Patient Reported Sleep Quality | 3 months
  Using questionnaire to evaluate patient satisfaction with sleep and associated symptoms. Scale will be subjective 1-10

SECONDARY OUTCOMES:
Sleep Data | 3 months
  Objective metrics collected via wearable sleep tracker - heart rate measured in BPM
Sleep Data | 3 months
  Objective metrics collected via wearable sleep tracker - heart rate variability measured in ms

IPD SHARING:
Plan to Share IPD: No